CLINICAL TRIAL: NCT07060885
Title: A Randomised Double-blind Placebo-controlled Phase III Field Trial Evaluating the Efficacy and Safety of the House Dust Mite (HDM) SLIT-tablet in Chinese Participants Aged 12-65 Years With HDM Allergic Rhinitis/Rhinoconjunctivitis With or Without Asthma
Brief Title: A Research Study of House Dust Mite (HDM) SLIT-tablet for the Treatment of HDM Allergy in Chinese Participants Aged 12-65
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-21; 2025-000321-14 (EudraCT Number)
Record Dates: First submitted 2025-07-01; First posted 2025-07-11 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-07

CONDITIONS: Allergic Rhinoconjunctivitis; Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active treatment (Experimental): HDM SLIT-tablet plus symptom-relieving medication used to alleviate allergic rhinitis/rhinoconjunctivitis symptoms.
  Interventions: Biological: HDM SLIT-tablet (12 SQ-HDM)
- Placebo (Placebo Comparator): Placebo sublingual tablet plus symptom-relieving medication used to alleviate allergic rhinitis/rhinoconjunctivitis symptoms.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: HDM SLIT-tablet (12 SQ-HDM) — For daily administration (1 tablet per day)
  Other Names: Acarizax, Odactra
  Arms: Active treatment
Other: Placebo — For daily administration (1 tablet per day)
  Arms: Placebo

SUMMARY:
A research study of house dust mite (HDM) SLIT-tablet for the treatment of HDM allergy in Chinese participants aged 12-65.

DETAILED DESCRIPTION:
The trial aims to evaluate efficacy of the house dust mite (HDM) SLIT-tablet compared to placebo in Chinese participants aged 12-65 with HDM allergic rhinitis/rhinoconjunctivitis with or without asthma. Efficacy will be assessed based on the total combined rhinitis score during the last 4 weeks of treatment.

The trial is a randomised, double-blind, parallel-group, placebo-controlled, multi-site, phase III trial conducted in China. The treatment period will be 24-28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Chinese subjects aged 12-65 years
* A clinical history of HDM AR/C (Allergic rhinitis/rhinoconjunctivitis) (with or without asthma) and with allergic rhinitis symptoms despite having received allergy pharmacotherapy during the previous year prior to screening
* Have a certain level of AR (Allergic rhinitis) symptoms on at least 8 of the last 14 days of the baseline period
* Use symptomatic medication for treatment of HDM allergic rhinitis during at least 8 of the last 14 days of the baseline period
* Positive skin prick test (SPT) and IgE (Immunoglobulin E) to D. pteronyssinus or D. farinae at screening
* Lung function ≥ 70% of predicted value

Exclusion Criteria:

* Sensitised and regularly exposed to perennial allergens
* Any nasal or pharyngeal condition that could interfere with the safety or efficacy evaluation
* Asthma requiring treatment with high dose of inhaled corticosteroid
* A relevant history of systemic allergic reaction

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Average daily total combined rhinitis score (TCRS) during the primary efficacy assessment period. | 4 weeks (primary efficacy assessment period), starting 24 weeks after initiation of IMP.
  The average daily TCRS evaluates the treatment effect as the difference in daily rhinitis symptoms and medication score (on a scale from 0-24) between participants treated with 12 SQ-HDM and placebo. Higher scores indicate more severe symptoms and/or more use of rhinitis medication. The endpoint is calculated as the average score of all reported daily values during the 4-week primary efficacy assessment period.

SECONDARY OUTCOMES:
Average daily values for rhinitis daily symptom score (DSS) during primary efficacy period. | 4 weeks (primary efficacy assessment period), starting 24 weeks after initiation of IMP.
  The average rhinitis DSS evaluates the treatment effect as the difference in daily rhinitis symptoms score (on a scale from 0-12) between participants treated with 12 SQ-HDM and placebo. Higher scores indicate more severe symptoms. The endpoint is calculated as the average score of all reported daily values during the 4-week primary efficacy assessment period.
Average daily values for rhinitis daily medication score (DMS) during primary efficacy period. | 4 weeks (primary efficacy assessment period), starting 24 weeks after initiation of IMP.
  Average rhinitis DMS evaluates the treatment effect as the difference in daily rhinitis medication use (on a scale of 0-12) between participants treated with 12 SQ-HDM and placebo. Higher scores indicate more medication use. The endpoint is calculated as the average score of all reported daily values during the 4-week primary efficacy assessment period.
Average daily total combined score (TCS) during primary efficacy period. | 4 weeks (primary efficacy assessment period), starting 24 weeks after initiation of IMP.
  Average rhinoconjunctivitis TCS evaluates the treatment effect as the difference in daily rhinoconjunctivitis symptoms and medication use (on a scale of 0-38) between participants treated with 12 SQ-HDM and placebo. Higher scores indicate more severe symptoms and/or more medication use. The endpoint is calculated as the average score of all reported daily values during the 4-week primary efficacy assessment period.
Average rhinoconjunctivitis DSS during the primary efficacy assessment period | 4 weeks (primary efficacy assessment period), starting 24 weeks after initiation of IMP.
  The average rhinoconjunctivitis DSS evaluates the treatment effect as the difference in daily rhinoconjunctivitis symptom score (on a scale of 0-18) between participants treated with 12 SQ-HDM and placebo. Higher scores indicate more severe symptoms. The endpoint is calculated as the average score of all reported daily values during the 4-week primary efficacy assessment period.
Average rhinoconjunctivitis DMS during the primary efficacy assessment period | 4 weeks (primary efficacy assessment period), starting 24 weeks after initiation of IMP.
  The average rhinoconjunctivitis DMS evaluates the treatment effect as the difference in daily rhinoconjunctivitis medication use (on a scale of 0-20) between participants treated with 12 SQ-HDM and placebo. Higher scores indicate more medication use. The endpoint is calculated as the average score of all reported daily values during the 4-week primary efficacy assessment period.

CONTACTS AND LOCATIONS:
Locations (30):
- China (30):
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - The first hospital affiliated Fujian medical University, Fuzhou, Fujian
  - The first affiliated hospital of guangzhou medical university-respiratory department, Guangzhou, Guangdong
  - The Third Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Third Affilliated Hospital of Southern Medical University, Guangzhou, Guangdong
  - Shenzhen Children's Hospital - Respiratory, Shenzhen, Guangdong
  - Huazhong University of science and Technology Union Shenzhen Hospital(Nanshan Hospital) - Endocrinology, Shenzhen, Guangdong
  - The Fifth Affiliated Hospital of Sun Yat-Sen University - University Hospital, Zhuhai, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The People's Hospital of Guangxi Zhuang Autonomous Region - Nephrology - Oncology, Nanning, Guangxi
  - Hainan General Hospital - Respiratory, Haikou, Hainan
  - The Third Hospital of Changsha - Pulmonology, Changshacun, Henan
  - The First Affiliated Hospital of University of South China - Endocrinology, Hengyang, Henan
  - Jingzhou Central Hospital - Otorhinolaryngology, Jingzhou, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology - Oncology, Wuhan, Hubei
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - Jiangsu Province Hospital/ The First Affiliated Hospital with Nanjing Medical University - Otorhinolaryngology, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University - Respiratory, Suzhou, Jiangsu
  - Nanchang University - The First Affiliated Hospital, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Xi an Jiaotong University (Xibei Hospital) - Nephrology, Xi'an, Shaanxi
  - Shanghai Jiaotong University School of Medicine, Ruijin Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Peking Union Medical College Hospital, Beijing, Sichuan
  - Sichuan University - West China Second University Hospital (WCSUH) (West China Women's and Children's Hospital), Chengdu, Sichuan
  - West China Hospital of Sichuan University - Otorhinolaryngology, Chengdu, Sichuan
  - The First Affiliated Hospital of Chongqing Medical University - Respiratory, Chongqing, Sichuan
  - Zhejiang provincial people's hospital, Hangzhou, Zhejiang
  - The 2nd School of Medicine, WMU/The 2nd Affiliated Hospital and Yuying Children's Hospital of WMU - Pediatrics, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No